CLINICAL TRIAL: NCT02998424
Title: Pupillary Diameter Without Stimulation Under Different Concentrations of Propofol Alone
Brief Title: Pupillary Diameter Under Different Concentrations of Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PD and propofol
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia
Keywords: propofol; pupillary diameter
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol 1 µg/ml (Experimental): Patients received a propofol infusion at an effect-site concentration of 1 µg/ml at the beginning of induction of general anesthesia for elective surgery.
  Pupillary diameter measurement after 10 minutes.
  Interventions: Drug: Propofol; Device: Pupillary diameter measurement
- Propofol 2 µg/ml (Experimental): Patients received a propofol infusion at an effect-site concentration of 2 µg/ml at the beginning of induction of general anesthesia for elective surgery.
  Pupillary diameter measurement after 10 minutes.
  Interventions: Drug: Propofol; Device: Pupillary diameter measurement
- Propofol 3 µg/ml (Experimental): Patients received a propofol infusion at an effect-site concentration of 3 µg/ml at the beginning of induction of general anesthesia for elective surgery.
  Pupillary diameter measurement after 10 minutes.
  Interventions: Drug: Propofol; Device: Pupillary diameter measurement

INTERVENTIONS:
Drug: Propofol — Continuous infusion
Device: Pupillary diameter measurement — Instantaneous measure

SUMMARY:
Resting pupillary diameter was measured at a randomized Effect-site target concentration of propofol used as a sole anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* patient who has reached puberty
* ASA I or II who is scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* neurologic, metabolic, ocular disease
* chronic pain
* under medication that interferes with autonomic nervous system
* obesity
* patient requiering a rapid sequence induction

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pupillary diameter | Instantaneous measure, 10 minutes after the beginning of the study period

SECONDARY OUTCOMES:
Bispectral Index (BIS) | continuous measure, recorded10 minutes after the beginning of the study period
Heart rate | continuous measure, recorded10 minutes after the beginning of the study period
Observer's Assessment of Alertness/Sedation Scale (OAAS) | 10 minutes after the beginning of the study
  Clinical score

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, MD-PHD, Study Director — Hopital Armand Trousseau, Université Paris 6, Département d'anesthésie
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabourdin N, Meniolle F, Chemam S, Rigouzzo A, Hamza J, Louvet N, Constant I. Effect of Different Concentrations of Propofol Used as a Sole Anesthetic on Pupillary Diameter: A Randomized Trial. Anesth Analg. 2020 Aug;131(2):510-517. doi: 10.1213/ANE.0000000000004362. PMID 31490817